CLINICAL TRIAL: NCT05309135
Title: A Phase 1, Double-Masked, Randomized, Safety and Efficacy, Single Center Clinical Evaluation of Corneal Injection for Endothelial Dysfunction Using Human Corneal Endothelial Cell Therapy (HCEC-1) in Adult Subjects With Corneal Edema Secondary to Endothelial Dysfunction
Brief Title: A Safety and Efficacy Study of Corneal Injection for Endothelial Dysfunction Using Human Corneal Endothelial Cell Therapy in Subjects With Corneal Edema Secondary to Endothelial Dysfunction
Acronym: Escalon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aurion Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-HCEC-1-004
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Corneal Edema
MeSH Terms: conditions — Corneal Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Within the treated groups, the sponsor, investigator, assessor, and subject will be masked to the assigned dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose Rho kinase inhibitor Y-27632 (Active Comparator): Low dose Rho kinase inhibitor Y-27632
  Interventions: Drug: HCEC-1
- Mid dose Rho kinase inhibitor Y-27632 (Active Comparator): Mid dose Rho kinase inhibitor Y-27632
  Interventions: Drug: HCEC-1
- High dose Rho kinase inhibitor Y-27632 (Active Comparator): High dose Rho kinase inhibitor Y-27632
  Interventions: Drug: HCEC-1

INTERVENTIONS:
Drug: HCEC-1 — HCEC-1 = human cultured corneal endothelial cells and Rho kinase Y-27632 inhibitor

SUMMARY:
The purpose of this study is to assess the safety of a fixed dose of human corneal endothelial cells when administered with varying concentrations of Rho kinase inhibitor (Y-27632) in patients with corneal edema secondary to endothelial dysfunction.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have given written informed consent (signed and dated by subject or legal guardian), and any authorizations required by local law and be able to comply with all study requirements
2. Clinical diagnosis of corneal edema secondary to endothelial dysfunction
3. Best Corrected Visual Acuity (BCVA) no worse than 20/800 ETDRS (1.6 LogMAR) or better than 20/63 (0.5 LogMAR) in the study eye

Key Exclusion Criteria:

1. Keratoconus or other conditions of corneal thinning/ectasia
2. Progressive stromal or anterior corneal dystrophies
3. Pre-operative corneal epithelial, sub-epithelial or stromal staining, scarring or other opacity that is paracentral/central and visually significant, but not suspected to be secondary to corneal endothelial disease with the potential to improve from treatment with HCEC-1
4. Prior ophthalmic surgery including cataract surgery except as noted above in Inclusion Criterion #4, corneal transplantation, glaucoma (MIGS, iridectomy, trabeculectomy, valve), or vitreo-retinal surgery, aphakia, anterior chamber-IOL or iris claw IOL, multifocal IOL.
5. Relative Afferent Pupillary Defect (RAPD) in the study eye
6. Uncontrolled glaucoma or an IOP greater than 24 mmHg that is not controlled with topical beta blockers alone at the time of the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment Emergent Ocular Adverse Events (TEAEs) | 12 months
Incidence and severity of non-ocular TEAEs | 12 months

SECONDARY OUTCOMES:
Change from baseline in Central Corneal Thickness (CCT) as measured by pachymetry | 12 months
Change from baseline in Best-Corrected Visual Acuity (BCVA) as measured by LogMAR score | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Site, San Salvador, El Salvador

IPD SHARING:
Plan to Share IPD: No
The study plan and protocol will be shared with the study center and other researchers per request.